CLINICAL TRIAL: NCT03378427
Title: Prospective Cohort Study on Patients With Tedizolid Prolonged Therapy for Orthopedic Device Infections
Brief Title: Tedizolid Prolonged Treatment for Prosthetic Joint Infections
Acronym: TEDIZOAM
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Tourcoing Hospital (Other)
Collaborators: Eric SENNEVILLE M.D. Ph.D. (Unknown)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2017-001238-24
Record Dates: First submitted 2017-10-24; First posted 2017-12-19 (Actual); Last update posted 2021-09-08 (Actual); Status verified 2020-04

CONDITIONS: Prosthetic Joint Infection
Keywords: Tedizolid; Adverse effects; Efficacy; prosthetic joint infection
MeSH Terms: interventions — tedizolid phosphate; Rifampin; Ofloxacin; Levofloxacin; Fusidic Acid; Clindamycin; Teicoplanin; Ciprofloxacin; Trimethoprim, Sulfamethoxazole Drug Combination; Doxycycline; Minocycline

STUDY DESIGN:
Intervention Model Description: Pilot study
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- Tedizolid Phosphate 200 MG [Sivextro] (Experimental): All included patients will receive prolonged (>= 6 weeks) tedizolid treatment given orally.
  Interventions: Drug: Tedizolid Phosphate 200 MG [Sivextro]

INTERVENTIONS:
Drug: Tedizolid Phosphate 200 MG [Sivextro] — Antibiotic treatment (monotherapy or combination) targeting bacteria cultured from per operative samples.
  Other Names: rifampin; ofloxacin; levofloxacin; fusidic acid; clindamycin; teicoplanin; ciprofloxacin; trimethoprim-sulfamethoxazole; doxycycline; minocycline

SUMMARY:
Pilot study the aim of which is to obtain reliable data on the tolerance, compliance and efficacy of Tedizolid used as prolonged (≥ 6 weeks) monotherapy or in combination therapy for the treatment of patients with orthopedic device infections due to Gram positive cocci.

DETAILED DESCRIPTION:
Background: The antibiotic treatment of patients with orthopedic device infections (e.g. prosthetic joint and osteosynthesis) is limited by the tolerance of prolonged administration of antibiotics and the high level of antibiotic resistance of some pathogens.

The prolonged intravenous administration of antibiotics exposes the patients to the occurrence of adverse events and it is generally recommended to favor oral treatment provided high oral bioavailable agents can be used with regard to the patient's characteristics and the antibiotic susceptibility profile of the pathogens.

Gram positive cocci especially coagulase negative staphylococci (CoNS) are predominant bacteria responsible for orthopedic device infections. The use of the oxazolidinone agent Linezolid in these settings has been validated by some studies in particular in combination with Rifampin but both hematologic, neurologic and metabolic potential toxicity limits treatment durations of more than two to three weeks. The risk of drug-drug interaction with any product having a mono-amine-oxydase inhibitor (MAOI) activity is another limiting problem with Linezolid use.

In addition, the wide use of Linezolid has resulted in the emergence of CoNS carrying cfr genes responsible for high levels of Linezolid resistance. This is unfortunate as in many cases there is almost no other alternative for the oral treatment of orthopedic device infections due to these strains.

Tedizolid intrinsic properties may improve the oxazolidinone treatment long term safety. Plus tedizolid should be active on CoNS strains resistant to linezolid.

Objectives: Obtain reliable data on the tolerance, compliance and efficacy of Tedizolid used as prolonged (≥ 6 weeks) monotherapy or in combination therapy for the treatment of patients with orthopedic device infections due to Gram positive cocci.

Hypothesis: As no data are currently available on long term safety of Tedizolid treatment, the investigators will compare the results of the present study regarding tolerance and efficacy with those of a historical cohort of comparable patients from our cohorts treated with Linezolid monotherapy or combination therapy for equivalent indications (data published in Journal of Antimicrobial Chemotherapy Legout L et al..2010).

Study Design: Prospective multicenter cohort study.

The objectives of the study are :

(i) to assess the tolerance of TEDIZOLID determined by the proportion of patients who experienced any adverse event attributable to TEDIZOLID during treatment and during 6 weeks after the antibiotic treatment, and (ii) to assess the efficacy of TEDIZOLID as single agent treatment or combined therapy for orthopedic infections due to TEDIZOLID susceptible bacteria determined by the proportion of patient with remission of the infection (i.e. absence of any local and systemic sign of infection in relation with the initial infection, any surgery for an infectious reason at the initial site or death related to the initial infection) determined one year after the end of the antibiotic treatment.

Microbiologic data from failure cases will be recorded in order to assess the presence of Tedizolid-resistant strains, relapsing infections, or superinfection.

Treatment: Tedizolid 200 mg once a day, administered orally for the entire treatment will be prescribed in patients after the definite culture results of peroperative samples will be available.

Daily doses of the antibiotics associated with tedizolid will be at the discretion of the clinician and will have to follow the institutional therapeutical protocols.

ELIGIBILITY:
Inclusion Criteria:

* Patient at least 18 years;
* Orthopedic device infection defined according to the French recommendations published in 2009 (Med Mal Infect 2009; 39:745-774) for which TEDIZOLID treatment is proposed according to the investigator's decision;
* Bacterial documentation of the infection will only be based on the results of reliable samples such as joint aspiration and peroperative samples.
* Requiring TEDIZOLID administration as a single antibiotic therapy or in combination therapy including another agent with proven activity against the involved pathogen(s);
* No contraindication to TEDIZOLID;
* Provide a signed informed consent for the trial.

Exclusion Criteria:

* pregnant women or of childbearing age without contraception, breastfeeding,
* intolerance to TEDIZOLID;
* allergy to LINEZOLID;
* bactéria non susceptible to TEDIZOLID;
* patient with uncertainty regarding the possibility to achieve one-year follow-up after the end of treatment.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 35 (Actual)
Dates: Start 2018-08-28 (Actual); Primary Completion 2020-10-22 (Actual); Study Completion 2021-08-22 (Actual)

PRIMARY OUTCOMES:
Bone marrow toxicity | From date of inclusion until 12 months after the end of treatment
  assessed on the values of hemoglobin, leucocytes, neutrophils and platelets counts, will be collected to determine the number of adverse event likely to be related to tedizolid treatment.
Peripheral neuropathy | From date of inclusion until 12 months after the end of treatment
  Paresthesia, dysesthesia, hypoesthesia, allodynia (confirmed by EMG examination), will be collected to determine the number of adverse event likely to be related to tedizolid treatment.
Metabolic acidosis | From date of inclusion until 12 months after the end of treatment
  dyspnea of unknown origin ; pH < 7.35 ; [ HCO3- ] < 22 mmol/L ; paCO2 < 45 mmHg ; lactates > 2 mmol/L, will be collected to determine the number of adverse event likely to be related to tedizolid treatment.
Serotoninergic syndrome | From date of inclusion until 12 months after the end of treatment
  will be collected to determine the number of adverse event likely to be related to tedizolid treatment.
Retrobulbar optic nevritis | From date of inclusion until 12 months after the end of treatment
  will be collected to determine the number of adverse event likely to be related to tedizolid treatment.

CONTACTS AND LOCATIONS:
Overall Officials: Eric SENNEVILLE, M.D. Ph. D., Study Chair — G. Dron Hospital, Tourcoing, France
Locations (2):
- France (2):
  - Hôpital Ambroise Paré, Boulogne-Billancourt
  - Hôpital de la Croix Rousse, Lyon

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Titecat M, Senneville E, Wallet F, Dezeque H, Migaud H, Courcol RJ, Loiez C. Microbiologic profile of Staphylococci isolated from osteoarticular infections: evolution over ten years. Surg Infect (Larchmt). 2015 Feb;16(1):77-83. doi: 10.1089/sur.2013.258. Epub 2015 Feb 4. PMID 25650692
- [Result] Titecat M, Senneville E, Wallet F, Dezeque H, Migaud H, Courcol RJ, Loiez C. Bacterial epidemiology of osteoarticular infections in a referent center: 10-year study. Orthop Traumatol Surg Res. 2013 Oct;99(6):653-8. doi: 10.1016/j.otsr.2013.02.011. Epub 2013 Aug 27. PMID 23988422
- [Result] Pulcini C, Couadau T, Bernard E, Lorthat-Jacob A, Bauer T, Cua E, Mondain V, Chichmanian RM, Dellamonica P, Roger PM. Adverse effects of parenteral antimicrobial therapy for chronic bone infections. Eur J Clin Microbiol Infect Dis. 2008 Dec;27(12):1227-32. doi: 10.1007/s10096-008-0570-y. Epub 2008 Sep 26. PMID 18818959
- [Result] Spellberg B, Lipsky BA. Systemic antibiotic therapy for chronic osteomyelitis in adults. Clin Infect Dis. 2012 Feb 1;54(3):393-407. doi: 10.1093/cid/cir842. Epub 2011 Dec 12. PMID 22157324
- [Result] Morata L, Tornero E, Martinez-Pastor JC, Garcia-Ramiro S, Mensa J, Soriano A. Clinical experience with linezolid for the treatment of orthopaedic implant infections. J Antimicrob Chemother. 2014 Sep;69 Suppl 1:i47-52. doi: 10.1093/jac/dku252. PMID 25135090
- [Result] Morata L, Senneville E, Bernard L, Nguyen S, Buzele R, Druon J, Tornero E, Mensa J, Soriano A. A Retrospective Review of the Clinical Experience of Linezolid with or Without Rifampicin in Prosthetic Joint Infections Treated with Debridement and Implant Retention. Infect Dis Ther. 2014 Dec;3(2):235-43. doi: 10.1007/s40121-014-0032-z. Epub 2014 Aug 20. PMID 25139552
- [Result] Senneville E, Legout L, Valette M, Yazdanpanah Y, Beltrand E, Caillaux M, Migaud H, Mouton Y. Effectiveness and tolerability of prolonged linezolid treatment for chronic osteomyelitis: a retrospective study. Clin Ther. 2006 Aug;28(8):1155-1163. doi: 10.1016/j.clinthera.2006.08.001. PMID 16982292
- [Result] Senneville E, Legout L, Valette M, Yazdanpanah Y, Giraud F, Beltrand E, Obert G, Dubreuil L, Migaud H, Mouton Y. Risk factors for anaemia in patients on prolonged linezolid therapy for chronic osteomyelitis: a case-control study. J Antimicrob Chemother. 2004 Oct;54(4):798-802. doi: 10.1093/jac/dkh409. Epub 2004 Aug 25. PMID 15329363
- [Result] Legout L, Senneville E, Gomel JJ, Yazdanpanah Y, Mouton Y. Linezolid-induced neuropathy. Clin Infect Dis. 2004 Mar 1;38(5):767-8. doi: 10.1086/381762. No abstract available. PMID 14986270
- [Result] Legout L, Valette M, Dezeque H, Nguyen S, Lemaire X, Loiez C, Caillaux M, Beltrand E, Dubreuil L, Yazdanpanah Y, Migaud H, Senneville E. Tolerability of prolonged linezolid therapy in bone and joint infection: protective effect of rifampicin on the occurrence of anaemia? J Antimicrob Chemother. 2010 Oct;65(10):2224-30. doi: 10.1093/jac/dkq281. Epub 2010 Jul 29. PMID 20675299
- [Result] Betriu C, Morales G, Rodriguez-Avial I, Culebras E, Gomez M, Lopez-Fabal F, Picazo JJ. Comparative activities of TR-700 (torezolid) against staphylococcal blood isolates collected in Spain. Antimicrob Agents Chemother. 2010 May;54(5):2212-5. doi: 10.1128/AAC.01653-09. Epub 2010 Feb 22. PMID 20176900
- [Result] Douros A, Grabowski K, Stahlmann R. Drug-drug interactions and safety of linezolid, tedizolid, and other oxazolidinones. Expert Opin Drug Metab Toxicol. 2015;11(12):1849-59. doi: 10.1517/17425255.2015.1098617. Epub 2015 Oct 12. PMID 26457865
- [Result] Flanagan SD, Bien PA, Munoz KA, Minassian SL, Prokocimer PG. Pharmacokinetics of tedizolid following oral administration: single and multiple dose, effect of food, and comparison of two solid forms of the prodrug. Pharmacotherapy. 2014 Mar;34(3):240-50. doi: 10.1002/phar.1337. Epub 2013 Aug 7. PMID 23926058
- [Result] Flanagan S, McKee EE, Das D, Tulkens PM, Hosako H, Fiedler-Kelly J, Passarell J, Radovsky A, Prokocimer P. Nonclinical and pharmacokinetic assessments to evaluate the potential of tedizolid and linezolid to affect mitochondrial function. Antimicrob Agents Chemother. 2015 Jan;59(1):178-85. doi: 10.1128/AAC.03684-14. Epub 2014 Oct 20. PMID 25331703
- [Result] Lodise TP, Bidell MR, Flanagan SD, Zasowski EJ, Minassian SL, Prokocimer P. Characterization of the haematological profile of 21 days of tedizolid in healthy subjects. J Antimicrob Chemother. 2016 Sep;71(9):2553-8. doi: 10.1093/jac/dkw206. Epub 2016 Jun 17. PMID 27317442
- [Result] Schmidt-Malan SM, Greenwood Quaintance KE, Karau MJ, Patel R. In vitro activity of tedizolid against staphylococci isolated from prosthetic joint infections. Diagn Microbiol Infect Dis. 2016 May;85(1):77-9. doi: 10.1016/j.diagmicrobio.2016.01.008. Epub 2016 Jan 12. PMID 26906190
- [Result] Morata L, Mensa J, Soriano A. New antibiotics against gram-positives: present and future indications. Curr Opin Pharmacol. 2015 Oct;24:45-51. doi: 10.1016/j.coph.2015.07.004. Epub 2015 Jul 30. PMID 26232669